CLINICAL TRIAL: NCT00905398
Title: Estudo da eficácia do Nilotinibe Concomitante à Quimioterapia no Tratamento de Pacientes Com Leucemia linfoblástica Aguda Filadélfia Positiva recém-diagnosticada
Brief Title: Nilotinib With Chemotherapy for the Treatment of Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia
Acronym: ALLPhi
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to excessive toxicity and low compliance to the protocol scheme.
Sponsor: Rony Schaffel (Other)
Responsible Party: Sponsor-Investigator, Rony Schaffel, MD, PhD, Universidade Federal do Rio de Janeiro
Organization: Universidade Federal do Rio de Janeiro (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrALL 01-08; ANVISA; 25351732040200851
Record Dates: First submitted 2009-05-15; First posted 2009-05-20 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Acute Lymphoblastic Leukemia
Keywords: Leukemia; Lymphoblastic; Acute; Philadelphia; BCR-ABL; Nilotinib; Treatment
MeSH Terms: conditions — Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nilotinib (Experimental): single arm study
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — 400mg, Oral, Bid, Daily for three years
  Other Names: Tasigna; AMN107

SUMMARY:
Patients with acute lymphoblastic leukemia and positivity for the breakpoint cluster region-Abelson murine leukemia (BCR-ABL) protein or the Philadelphia chromosome have a poor prognosis with standard chemotherapy. The prognosis seemed to improve following the adition of imatinibe, a BCR-ABL inhibitor, to the treatment but still a substantial amount of patients relapse or progress during treatment.

Nilotinib is a BCR-ABL inhibitor more potent than imatinib. It has been shown to be effective against most of the cells that bear mutations of the BCR-ABL protein leading to resistance to imatinibe.

The investigators' hypothesis is that the addition of nilotinib to a standard chemotherapy for acute lymphoblastic leukemia (ALL) will translate into more rapid BCR-ABL reduction and effectiveness against imatinib-resistant clones leading to less relapses and better survival.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Acute Lymphoblastic Leukemia (ALL)
* BCR-ABL positive positive by PCR (central Lab)
* No previous treatment for ALL except for corticoids and cyclophosphamide less than 600 mg/m2
* Must be able to swallow tablets
* Lab results within normal limits (Potassium, Calcium, Magnesio, Phosphorus, Transaminases, Alkaline Phosphatase, Bilirrubine, Amylase, Lypase)

Exclusion Criteria:

* Heart disease
* Interval QTc Fridericia > 480 msec
* Coumadin use
* Pregnancy
* PS = 4
* Previous medical history of etilism or/and pancreatic disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-05; Primary Completion 2012-06 (Actual); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Complete remission | Day + 21 and Day + 41

SECONDARY OUTCOMES:
Overall Survival | Three years
Molecular remission | Every three months until three years
Toxicity | Three times a week for the first 40 days than once weekly for the next 9 months than monthly for the next 2.1 years

CONTACTS AND LOCATIONS:
Overall Officials: Rony Schaffel, MD, PHD, Principal Investigator — Rio de Janeiro Federal University; Nelson Spector, MD, PHD, Study Chair — Rio de Janeiro Federal University; Belinda Simões, MD, PHD, Principal Investigator — São Paulo University (Ribeirão Preto)